CLINICAL TRIAL: NCT00358462
Title: Mycoplasma Genitalium Antibiotic Susceptibility and Treatment: A Randomized Double-blind Trial of the Efficacy of Azithromycin and Doxycycline for Clinical and Microbiological Cure of M. Genitalium in Men With Nongonococcal Urethritis
Brief Title: Mycoplasma Genitalium Antibiotic Susceptibility and Treatment (MEGA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Lisa Manhart, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26995; 05-0143 (protocol number) (Other: University of Washington); U19AI031448 (NIH); R01AI072728 (NIH)
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Urethritis
Keywords: NGU, M genitalium, Ureaplasma, azithromycin, doxycycline
MeSH Terms: conditions — Urethritis | interventions — Azithromycin; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active azithromycin+placebo doxycycline (Active Comparator): Active azithromycin (1g) and placebo doxycycline
  Interventions: Drug: Azithromycin
- Active doxycycline+placebo azithromycin (Active Comparator): Active doxycycline and placebo azithromycin
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Azithromycin — two 500mg tablets or four 250mg tablets administered as a single dose
  Other Names: Zithromax; Zmax
  Arms: Active azithromycin+placebo doxycycline
Drug: Doxycycline — one 100mg capsule administered twice daily for seven days
  Other Names: Doryx; Doxychel; Monodox; Oracea; Periostat; Vibra-Tabs; Vibramycin
  Arms: Active doxycycline+placebo azithromycin

SUMMARY:
The purpose of this study is to find out which of 2 different antibiotics, doxycycline or azithromycin, works best against germs that may cause nongonococcal urethritis.

Study participants will include approximately 1200 men, 16 years of age or older, attending a sexually transmitted diseases clinic in Seattle, Washington with clinical signs of urethral inflammation (>=5PMNs/HPF on a Gram-stained slide prepared from urethral exudates and/or a visible urethral discharge upon examination).

Urine specimens will be collected and tested for Mycoplasma genitalium and Ureaplasmas. Each participant will receive a blinded packet of study medication. Participants will answer an enrollment questionnaire and will also receive a log to complete between visits to record information about treatment adherence, side effects, symptoms, and sexual activity. All subjects will be asked to return for evaluation 3 weeks after the initial clinic visit. Subjects who test positive for M. genitalium and/or Ureaplasmas at the initial clinic visit will also be asked to return for a third study visit, 6 weeks following the initial clinic visit. During follow-up visits, participants will answer a follow-up questionnaire and will be re-evaluated for signs of urethritis. Those who were initially positive for M. genitalium and/or Ureaplasmas will be re-tested for these organisms.

Study participants with signs and/or symptoms of urethritis or who test positive for M. genitalium or Ureaplasmas at the follow-up study visit will receive another blinded treatment packet containing the alternate medication. Those who require additional treatment at the 6-week visit will be asked to return for a fourth follow-up study visit at 9-10 weeks. Study participants who did not test positive for M. genitalium or Ureaplasmas at the initial clinic visit, but who continue to demonstrate signs and/or symptoms of infection at their single follow-up study visit will treated according to clinic standard of care (after the study clinician unblinds their randomly-assigned treatment regimen).

DETAILED DESCRIPTION:
OBJECTIVES

The primary objective of this study is to determine the relative effectiveness of azithromycin and doxycycline in eradicating Mycoplasma genitalium and Ureaplasmas among men with nongonococcal urethritis (NGU).

Secondary objectives of this study are to:

* determine the sensitivity of persisting organisms to azithromycin and doxycycline by performing minimum inhibitory concentration (MIC) testing
* determine the relationship between persistence/recurrence of clinical signs and persistent/recurrent detection of M. genitalium and Ureaplasmas among men with NGU treated with azithromycin or doxycycline, measured by follow-up clinical exams and repeated assays performed on specimens collected at follow-up study visits

STUDY DESCRIPTION

1200 men with NGU, ages 16 and older, will be enrolled in a randomized double-blinded treatment trial. Urine samples, oral swabs, and urethral swabs will be obtained from each subject at the initial clinic visit. Urine specimens will be tested for M. genitalium and Ureaplasma. Study participants will be randomly assigned to receive one of two pre-packaged treatments: active doxycycline plus placebo azithromycin or active azithromycin plus placebo doxycycline. Subjects will complete a questionnaire, and will be given a simple standardized log in which they will be asked to keep track of adherence to the study drug, record solicited adverse events, note when symptoms disappear and/or reappear, and document sexual activity between study visits.

Subjects who test positive for M. genitalium or Ureaplasmas at the initial clinic visit will be asked to return for at least two follow-up study visits: at approximately 3 and 6 weeks following the initial clinic visit. During follow-up visits, participants will answer a follow-up questionnaire and will be re-evaluated for signs of urethritis and re-tested for M. genitalium and Ureaplasmas. Study participants with signs and/or symptoms of urethritis or who test positive for M. genitalium or Ureaplasmas at the follow-up study visits will receive a blinded treatment packet containing the alternate medication, or will be offered open-label moxifloxacin if the alternate treatment regimen was administered at the prior follow-up study visit. If additional treatment is administered at the 6-week follow-up study visit, a fourth study visit will be scheduled to occur approximately 9 or 10 weeks following the initial clinic visit.

Study participants who were negative for M. genitalium and Ureaplasma at enrollment will be asked to return for evaluation for a single follow-up study visit, approximately 3 weeks after the initial clinic visit. At this visit they will complete the follow-up questionnaire and provide specimens for future testing.

ELIGIBILITY:
Inclusion Criteria:

* Has a visible urethral discharge or greater than or equal to 5 polymorphonuclear leukocytes (PMNs) per high power field on a Gram-stained slide of a urethral swab sample
* Possesses and is willing to disclose valid contact information for follow-up
* English-speaking
* Gives informed consent
* Exhibits understanding of study procedures
* Exhibits ability to comply with study procedures for the entire length of the study

Exclusion Criteria:

* Has previously participated in this study
* Has taken antibiotics within the prior month
* Has known allergies to tetracyclines or azithromycin
* Is being treated with any of the following: warfarin, ergot derivatives, pimozide (Orap), propafenone (Rytmonorm, Rythmol), disopyramide (Norpace, Rythmodan), rifampin, digoxin, isotretinoin, or methotrexate
* Has received a kidney, heart, or lung transplant.
* Is undertaking concomitant systemic steroid therapy

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2007-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Manhart, PhD, Principal Investigator — University of Washington
Locations (1):
- Public Health -- Seattle & King County Sexually Transmitted Diseases Clinic located at Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Khosropour CM, Manhart LE, Gillespie CW, Lowens MS, Golden MR, Jensen NL, Kenny GE, Totten PA. Efficacy of standard therapies against Ureaplasma species and persistence among men with non-gonococcal urethritis enrolled in a randomised controlled trial. Sex Transm Infect. 2015 Aug;91(5):308-13. doi: 10.1136/sextrans-2014-051859. Epub 2015 Jan 23. PMID 25616607
- [Derived] Khosropour CM, Manhart LE, Colombara DV, Gillespie CW, Lowens MS, Totten PA, Golden MR, Simoni J. Suboptimal adherence to doxycycline and treatment outcomes among men with non-gonococcal urethritis: a prospective cohort study. Sex Transm Infect. 2014 Feb;90(1):3-7. doi: 10.1136/sextrans-2013-051174. Epub 2013 Oct 8. PMID 24106340
- [Derived] Manhart LE, Gillespie CW, Lowens MS, Khosropour CM, Colombara DV, Golden MR, Hakhu NR, Thomas KK, Hughes JP, Jensen NL, Totten PA. Standard treatment regimens for nongonococcal urethritis have similar but declining cure rates: a randomized controlled trial. Clin Infect Dis. 2013 Apr;56(7):934-42. doi: 10.1093/cid/cis1022. Epub 2012 Dec 7. PMID 23223595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men were recruited from a sexually transmitted diseases clinic in Seattle, Washington from January 2007 to July 2011
Groups:
- Active Azithromycin + Placebo Doxycycline: Azithromycin : two 500mg tablets or four 250mg tablets administered as a single dose
- Active Doxycycline + Placebo Azithromycin: Doxycycline : one 100mg capsule administered twice daily for seven days
Period: Overall Study
Arm/Group | Active Azithromycin + Placebo Doxycycline | Active Doxycycline + Placebo Azithromycin
Started | 304 | 302
Completed | 245 | 238
Not Completed | 59 | 64

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Azithromycin + Placebo Doxycycline | Active Doxycycline + Placebo Azithromycin | Total
Number analyzed (Participants) | 304 | 302 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.8) | 33.3 (10.1) | 33.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 304 | 302 | 606
Region of Enrollment [Number; unit: participants]
  United States | 304 | 302 | 606

OUTCOME MEASURES:

1. Primary Outcome: mITT Analysis of Eradication of M. Genitalium at First Follow-up Study Visit
Description: Microbiologic cure of M. genitalium at first follow-up visit (defined as a negative in-house PCR test performed on urine)
Time Frame: approximately 3 weeks after initial study visit (allowable window is 2-5 weeks after initial study visit)
Population: mITT population (defined as urethral symptoms or visible discharge plus >=5PMNs/HPF at baseline) who tested positive for M. genitalium at baseline
Measure: Number; unit: participants
Arm/Group | Active Azithromycin + Placebo Doxycycline | Active Doxycycline + Placebo Azithromycin
Number analyzed (Participants) | 38 | 27
participants | 15 | 8

2. Primary Outcome: mITT Analysis of Eradication of U. Urealyticum at First Follow-up Visit
Description: Microbiologic cure, defined as negative PCR for U. urealyticum (if cultured), or negative culture at first follow-up visit
Time Frame: 3 weeks (allowable window 2-5)
Population: mITT population (defined as urethral symptoms or visible discharge plus >=5PMNs/HPF at baseline) who tested positive for U. urealyticum at baseline
Measure: Number; unit: participants
Arm/Group | Active Azithromycin + Placebo Doxycycline | Active Doxycycline + Placebo Azithromycin
Number analyzed (Participants) | 52 | 55
participants | 39 | 38

3. Secondary Outcome: Clinical Cure Among Case Subjects Who Were Positive for M. Genitalium at the Initial Study Visit
Description: Proportion of men with M. genitalium at the initial study visit who had clinical cure, defined as <5 PMNs/HPF (with or without urethral symptoms) on a urethral Gram stain and absence of urethral discharge at follow-up.
Time Frame: approximately 3 weeks after initial study visit (allowable window is 2-5 weeks after initial study visit)
Population: mITT population
Measure: Number; unit: participants
Arm/Group | Active Azithromycin+Placebo Doxycycline | Active Doxycycline+Placebo Azithromycin
Number analyzed (Participants) | 38 | 27
participants | 24 | 13

4. Secondary Outcome: Clinical Cure Among Case Subjects Who Were Positive for Ureaplasmas at the Initial Study Visit
Description: Proportion of men with Ureaplasma urealyticum at the initial study visit who had clinical cure, defined as <5 PMNs/HPF (with or without urethral symptoms) on a urethral Gram stain and absence of urethral discharge at follow-up.
Time Frame: approximately 3 weeks after initial study visit (allowable window is 2-5 weeks after initial study visit)
Population: mITT population
Measure: Number; unit: participants
Arm/Group | Active Azithromycin+Placebo Doxycycline | Active Doxycycline+Placebo Azithromycin
Number analyzed (Participants) | 52 | 55
participants | 43 | 40

5. Secondary Outcome: Minimum Inhibitory Concentrations (MIC) of M. Genitalium for Azithromycin
Description: In vitro susceptibiities of M. genitalium to azithromycin
Time Frame: baseline
Population: Participants with recovered isolates that successfully underwent in vitro assessment of antibiotic susceptibilities
Measure: Count of Participants; unit: Participants
Groups:
- Cultivated Isolates: Azithromycin MIC's
Arm/Group | Cultivated Isolates
Number analyzed (Participants) | 56
Participants
  MIC range <=0.001 - 0.004 ug/ml | 31
  MIC range >8 ug/ml | 25

6. Secondary Outcome: Minimum Inhibitory Concentrations (MIC) of M. Genitalium for Doxycycline
Description: In vitro susceptibilities of M. genitalium to doxycycline
Time Frame: baseline
Measure: Median (Full Range); unit: MIC (ug/mL)
Groups:
- Cultivated Isolates: Cultivated M. genitalium isolates that successfully underwent in vitro MICs for doxycycline
Arm/Group | Cultivated Isolates
Number analyzed (Participants) | 61
MIC (ug/mL) | 0.5 [0.125 to 2.0]

7. Secondary Outcome: Minimum Inhibitory Concentrations (MIC) of U. Ureaplasma Biovar 2
Description: In vitro susceptibilities of U. urealyticum biovar 2
Time Frame: baseline
Population: isolates
Measure: Median (Full Range); unit: MIC (ug/mL)
Groups:
- Azithromycin: Cultivated U. urealyticum biovar 2 isolates that successfully underwent in vitro MICs for azithromycin
- Doxycycline: Cultivated U. urealyticum biovar 2 isolates that successfully underwent in vitro MICs for doxycycliine
- Moxifloxacin: Cultivated U. urealyticum biovar 2 isolates that successfully underwent in vitro MICs for moxifloxacin
Arm/Group | Azithromycin | Doxycycline | Moxifloxacin
Number analyzed (Participants) | 22 | 22 | 22
MIC (ug/mL) | 1.00 [0.25 to 2.00] | 0.5 [0.125 to 1.00] | 0.5 [0.25 to 1.00]

8. Secondary Outcome: Minimum Inhibitory Concentrations (MIC) of U. Parvum
Description: In vitro susceptibilities of U. parvum
Time Frame: baseline
Population: isolates
Measure: Median (Full Range); unit: MIC (ug/mL)
Groups:
- Azithromycin: Cultivated U. parvum isolates that successfully underwent in vitro MICs for azithromycin
- Doxycycline: Cultivated U. parvum isolates that successfully underwent in vitro MICs for doxycycline
- Moxifloxacin: Cultivated U. parvum isolates that successfully underwent in vitro MICs for moxifloxacin
Arm/Group | Azithromycin | Doxycycline | Moxifloxacin
Number analyzed (Participants) | 8 | 8 | 8
MIC (ug/mL) | 0.5 [0.125 to 2.00] | 0.25 [0.125 to 0.50] | 0.25 [0.125 to 0.50]

ADVERSE EVENTS:
Arm/Group | Active Azithromycin + Placebo Doxycycline | Active Doxycycline + Placebo Azithromycin
Serious Adverse Events (participants affected / at risk) | 1/304 | 3/302
Other Adverse Events (participants affected / at risk) | 53/304 | 56/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Azithromycin + Placebo Doxycycline (N=304) | Active Doxycycline + Placebo Azithromycin (N=302)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Broken leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Unstable mental status (Psychiatric disorders) | 1 (1) | 0 (0)
Optic neuritis (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Azithromycin + Placebo Doxycycline (N=304) | Active Doxycycline + Placebo Azithromycin (N=302)
Nausea (Gastrointestinal disorders) | 28 (73) | 36 (68)
Diarrhea (Gastrointestinal disorders) | 31 (74) | 35 (47)
Vomiting (General disorders) | 6 (7) | 7 (7)
Rash (General disorders) | 6 (7) | 7 (7)
Other (Gastrointestinal disorders) | 12 (32) | 17 (32) — flu, cold, URTI; STD/genital injury or pain; dizziness; injuries; dry mouth; non-rash skin condition);elective medical procedure; mild bleeding; sunburn; tightness in head, neck

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No